CLINICAL TRIAL: NCT04613830
Title: Continuous Erector Spinae Plane Local Anesthetic Infusion for Postoperative Analgesia in Pediatric Patients Undergoing Nephrectomy: Randomized Controlled Study
Brief Title: Continuous Erector Spinae Block for Post Analgesia in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, Associated professor of anesthesia,ICU and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 515
Record Dates: First submitted 2020-10-23; First posted 2020-11-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Bupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erector spinae group (Active Comparator): patient will be placed in a sitting position under complete aseptic condition and a cover sheath will be used for the ultrasound probe with an appropriate amount of lubricating gel applied on the probe, a high-frequency linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the L3 spinous process. This should reveal three muscles superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae.
  Interventions: Drug: Bupivacaine Hydrochloride
- Opioid GROUP (Placebo Comparator): Patient in group T will intravenously administrate dose of 1 mg/kg/8hr tramal ( opioid) to be increased upon patient needs up to 2mg/kg/6hr as rescue analgesic.
  Interventions: Drug: Tramadol hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — The patient will be placed in a sitting position under complete aseptic condition and a cover sheath will be used for the ultrasound probe with an appropriate amount of lubricating gel applied on the probe, a high-frequency linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the L3 spinous process. This should reveal three muscles superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. then injecte bupivacaine hydrochloride
  Other Names: erector spinae block
  Arms: Erector spinae group
Drug: Tramadol hydrochloride — Patients in group Tramadol will intravenously administrate dose of 1 mg/kg/8hr tramal to be increased upon patient needs up to 2mg/kg/6hr as rescue analgesic
  Other Names: opioid group
  Arms: Opioid GROUP

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy of erector spinae plane block in pediatric cancer patients undergoing open nephrectomy

DETAILED DESCRIPTION:
* Sixty patients will be included in this prospective randomized study. The patients will be allocated into two groups: the ESPB group (group E, n = 30) and the tramal group (group T, n =30).
* All patients will receive standard general anesthesia. Ultrasound-guided ESPB will be performed to group erector spinae plane block

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA II.
* Patients (age 2-7yrs) scheduled for open nephrectomy for malignant kidney tumors

Exclusion Criteria:

* History of psychological disorders.

  * Known sensitivity or contraindication to local anesthetics.
  * Localized infection at the site of block.
  * patients with coagulopathy or an (INR ≥ 2)

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
total amount of opioid consumption in milligram | 48 hours
  total amount of opioid consumption in the frist 48hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: fatma el sherif, MD, Principal Investigator — Assiut University
Locations (1):
- South Egypt Cancer instIitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No